CLINICAL TRIAL: NCT07264257
Title: Choline and Brain Functioning in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: Balchem Corporation (Industry)
Responsible Party: Principal Investigator, Julie Dumas, Professor, University of Vermont
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: STU1720
Record Dates: First submitted 2025-09-10; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-09

CONDITIONS: Menopause
Keywords: cognition; fMRI; working memory; choline
MeSH Terms: interventions — Choline

STUDY DESIGN:
Intervention Model Description: placebo controlled study
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Choline (Experimental): Each subject completes two study days with choline and placebo.
  Interventions: Dietary Supplement: Choline
- Placebo (Experimental): Each subject completes two study days with choline and placebo.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Choline — Each subject gets one 1650 mg oral choline dose or placebo on each of two study days.
  Arms: Choline
Dietary Supplement: Placebo — Each subject gets one 1650 mg oral choline dose or placebo on each of two study days.
  Arms: Placebo

SUMMARY:
This study will use a randomized placebo-controlled trial to examine a single oral dose of 1650 mg choline influences brain functioning as measured by fMRI.

DETAILED DESCRIPTION:
Choline is an essential nutrient that, in addition to its role in the brain, has a number of critical structural and physiologic roles throughout the body, including providing structural integrity and signaling function for cell membranes, facilitating lipid transport from the liver, and acting as the major source of methyl groups through diet. Aside from dietary intake, the only source of choline in the body is de novo synthesis of phosphatidylcholine, catalyzed by phosphatdylethanolamine-N-methyltransferase (PEMT). The PEMT gene has several estrogen-responsive components in its promoter region and is induced by estrogen. Post-menopausal (hypo-estrogenic) women with loss of function mutations in PEMT have been found to exhibit end-organ damage typical of choline deficiency.

Choline is also involved in the synthesis of acetylcholine, a major neurotransmitter and the central and peripheral nervous systems. The relationship between brain effects of the normal functioning of the cholinergic system and hormone changes after menopause has been demonstrated in preclinical studies in rat models and in experimentally in human studies. While the preclinical and clinical experiment studies have many similar findings regarding the influence of estrogen on cholinergic functioning, what is not clear from this research is how individual differences arise in the effects of the hormone withdrawal after menopause on brain functioning in middle aged women. It is possible that the estrogen control of the transcription of the PEMT gene may influence the availability of choline.

This study will examine the effects of a single oral dose of oral dose of 1650 mg choline versus placebo in 20 healthy postmenopausal women aged 50-65 years. Choline or placebo will be administered three hours before an MRI session where subjects undergo functional MRI scans.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 50-65 years
* Postmenopausal: Women who are postmenopausal will have not had a period in the last 12 months, have FSH>30 IU/L, and estradiol (E2) <50 pg/ml.
* Nonsmokers
* Not taking hormone therapy, SSRIs, phytoestrogens, SERMS, or antiestrogen medications and will be at least one year without such treatment
* Physically healthy
* No cardiovascular disease other than mild hypertension. Subjects will also not have current untreated or unremitted Axis I or II psychiatric or cognitive disorders (see screening below).
* IQ in the normal range >80
* Normal neuropsychological test performance

Exclusion Criteria:

* MCI or dementia - Montreal Cognitive Assessment <26, Mattis Dementia Rating Scale <130, and Global Deterioration Scale >2
* History of cancer treatment with cytotoxic and/or ongoing (current) maintenance targeted chemotherapy
* Blood pressure > 160/100 (untreated)
* Untreated thyroid disease
* Significant cardiovascular disease
* Asthma or COPD
* Active peptic ulcer
* Hyperthyroidism
* Epilepsy
* Current untreated or unremitted Axis I psychiatric disorders
* Use of medications on the Prohibited medications (see list)

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
BOLD Signal during fMRI working memory task | Measured on each of the two study days
  fMRI BOLD signal during a working memory task

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Dumas, PhD, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: Yes
After data are published, deidentified data will be made available to those who request access.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: 10/2025 until 9/2030